CLINICAL TRIAL: NCT03215641
Title: Effect of Personal Activity Trackers on Weight Loss in Children Enrolled in a Comprehensive Behavioral Family Lifestyle Intervention (CBFLI) Program
Brief Title: Is it Helpful to Use Fitbits in a Family Based Weight Loss Program?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Academic Pediatric Association (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-15-00269; R25DK096944 (NIH)
Record Dates: First submitted 2016-05-20; First posted 2017-07-12 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Pediatric Obesity
Keywords: obesity; pediatrics; weight management program; Fitbit; personal activity tracker
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The control group families will participate in the standard Body Works weight loss program. They will fill out brief surveys regarding their physical activity on a weekly basis, but otherwise will receive the standard curriculum. they will receive weekly feedback based on their physical activity surveys.
- Intervention (Experimental): The intervention group families will be given fitbits on the first day of the Body Works program. They will otherwise receive the same curriculum as the control families. the will fill out the same physical activity surveys as the control families. they will receive weekly feedback based on the objectively measured physical activity.
  Interventions: Device: Fitbit

INTERVENTIONS:
Device: Fitbit — The Fitbit is a consumer-grade personal activity tracker. It is used to track physical activity. Patients will be given devices at the beginning of the study, and they will continue to use it for 7 weeks. Their data will be collected on a weekly basis, and patients will receive feedback on their level of activity based on the Fitbit data.
  Arms: Intervention

SUMMARY:
This study evaluates the role of personal activity trackers to help improve weight loss or weight maintenance for children and their parents enrolled in a comprehensive weight loss program.

DETAILED DESCRIPTION:
Childhood obesity rates have tripled in the last 30 years, with as many as 50% of children in the US being obese or overweight. High-intensity comprehensive behavioral family lifestyle intervention (CBFLI) programs have been shown to be among the most effective interventions for weight loss in children. However, these programs are time- and resource-intensive with high rates of recidivism. Personal activity trackers (PAT) provide objectively measured physical activity data and are more reliable than self-report. These devices can also have a motivational impact. The investigators intend to study the effects of these devices and their data on behavior change and weight loss for both parents and children enrolled in a CBFLI program. The investigators will objectively measure the level of activity of both members of the parent-child dyad, explore the relationship between parent-child activity levels and its effect on each other, as well as on overall weight loss or weight maintenance.

ELIGIBILITY:
Inclusion Criteria:

* All individuals enrolled in BodyWorks who are at least 7 years old meet inclusion criteria for this study. there is no maximum age for participation.

Exclusion Criteria:

Unable to wear PAT as described in study protocol Unwilling to wear PAT Unwilling to participate in the study

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-08; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
BMI-z score | Baseline to program completion (~8 weeks)
  change in BMI-z score

SECONDARY OUTCOMES:
Impact of fitbit on program attendance | Baseline to program completion (~8 weeks)
  The investigators will evaluate if families that receive fitbits attend more sessions (out of 7 total sessions) by recording their attendance at each session
impact of fitbit on program completion rate | Baseline to program completion (~8 weeks)
  The investigators will evaluate if families that receive fitbits complete the program at a higher rate (completion is defined as having attended at least 4 out of 7 sessions).

OTHER OUTCOMES:
relationship between change in child weight, in Kg, and daily parent steps taken as measured by the Fitbit | Baseline to program completion (~8 weeks
  evaluate whether parents who are more active have children who are more likely to lose weight

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Espinoza, MD, Principal Investigator — Children's Hospital Los Angeles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang G, Dietz WH. Economic burden of obesity in youths aged 6 to 17 years: 1979-1999. Pediatrics. 2002 May;109(5):E81-1. doi: 10.1542/peds.109.5.e81. PMID 11986487
- [Background] Janicke DM, Steele RG, Gayes LA, Lim CS, Clifford LM, Schneider EM, Carmody JK, Westen S. Systematic review and meta-analysis of comprehensive behavioral family lifestyle interventions addressing pediatric obesity. J Pediatr Psychol. 2014 Sep;39(8):809-25. doi: 10.1093/jpepsy/jsu023. Epub 2014 May 13. PMID 24824614
- [Background] Troiano RP, McClain JJ, Brychta RJ, Chen KY. Evolution of accelerometer methods for physical activity research. Br J Sports Med. 2014 Jul;48(13):1019-23. doi: 10.1136/bjsports-2014-093546. Epub 2014 Apr 29. PMID 24782483
- [Background] Buttitta M, Iliescu C, Rousseau A, Guerrien A. Quality of life in overweight and obese children and adolescents: a literature review. Qual Life Res. 2014 May;23(4):1117-39. doi: 10.1007/s11136-013-0568-5. Epub 2013 Nov 19. PMID 24249217
- [Background] Guinhouya BC, Samouda H, de Beaufort C. Level of physical activity among children and adolescents in Europe: a review of physical activity assessed objectively by accelerometry. Public Health. 2013 Apr;127(4):301-11. doi: 10.1016/j.puhe.2013.01.020. Epub 2013 Apr 10. PMID 23582270
- [Background] Lytle LA. Dealing with the childhood obesity epidemic: a public health approach. Abdom Imaging. 2012 Oct;37(5):719-24. doi: 10.1007/s00261-012-9861-y. PMID 22395212
- [Background] Trasande L, Elbel B. The economic burden placed on healthcare systems by childhood obesity. Expert Rev Pharmacoecon Outcomes Res. 2012 Feb;12(1):39-45. doi: 10.1586/erp.11.93. PMID 22280195
- [Background] Wilks DC, Besson H, Lindroos AK, Ekelund U. Objectively measured physical activity and obesity prevention in children, adolescents and adults: a systematic review of prospective studies. Obes Rev. 2011 May;12(5):e119-29. doi: 10.1111/j.1467-789X.2010.00775.x. PMID 20604868
- [Background] Whitlock EP, O'Connor EA, Williams SB, Beil TL, Lutz KW. Effectiveness of weight management interventions in children: a targeted systematic review for the USPSTF. Pediatrics. 2010 Feb;125(2):e396-418. doi: 10.1542/peds.2009-1955. Epub 2010 Jan 18. PMID 20083531
- [Background] Trasande L, Chatterjee S. The impact of obesity on health service utilization and costs in childhood. Obesity (Silver Spring). 2009 Sep;17(9):1749-54. doi: 10.1038/oby.2009.67. Epub 2009 Mar 19. PMID 19300433
- [Background] Oude Luttikhuis H, Baur L, Jansen H, Shrewsbury VA, O'Malley C, Stolk RP, Summerbell CD. Interventions for treating obesity in children. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD001872. doi: 10.1002/14651858.CD001872.pub2. PMID 19160202
- [Background] Finkelstein EA, Trogdon JG. Public health interventions for addressing childhood overweight: analysis of the business case. Am J Public Health. 2008 Mar;98(3):411-5. doi: 10.2105/AJPH.2007.114991. Epub 2008 Jan 30. PMID 18235061
- [Derived] Espinoza JC, Deavenport-Saman A, Solomon O, Chowdhuri S, Wee CP, Azen C, Orozco J, Kreutzer C, Yin L. Not just at school: Inclusion of children with autism spectrum disorder in a weight management program in a community pediatric setting. Autism. 2021 Apr;25(3):642-655. doi: 10.1177/1362361321993710. Epub 2021 Feb 24. PMID 33626921